CLINICAL TRIAL: NCT02919085
Title: Effect of Spontaneously Breathing Critical Patients Mobilization on Respiratory and Peripheral Muscle Strength and Functional Capacity.
Brief Title: Effect of Critical Patients Mobilization on Respiratory and Peripheral Muscle Strength and Functional Capacity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria Karoline de França Richtrmoc, Master student, Universidade Federal de Pernambuco
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01110031483
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Intensive Care Unit Syndrome; Muscle Weakness
MeSH Terms: conditions — Muscle Weakness | interventions — Early Ambulation

ARMS (1):
- Mobilization (Experimental)
  Interventions: Procedure: Early ambulation

INTERVENTIONS:
Procedure: Early ambulation — Procedure to accelerate the ability of a patient to walk or move about by reducing the time to ambulation. It is characterized by a shorter period of hospitalization or recumbency than is normally practiced.
  Other Names: Early mobilization

SUMMARY:
To analyze changes on respiratory muscle strength, peripheral and functional capacity of critically ill patients with clinical and surgical etiology, breathing spontaneously and bedridden, within 48 hours of admission to the intensive care unit (ICU) and if there are correlations among these variables. This is an observational study. Respiratory muscle strength will be assessed through the maximum inspiratory pressure (MIP) and maximal expiratory pressure (MEP) and peripheral muscle strength, by the Medical Research Council score (MRC) and hand grip test and functional capacity through the Functional Independence Measure (FIM) and Physical Function ICU Test Score (PFIT-s) in the period between 24h and 48h of hospitalization in the adult ICU. For descriptive purposes, the sample will be stratified according to clinical and surgical characteristics. Correlations will be determined using the Pearson test, with significance level of p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* Breathing spontaneously
* Length of stay in ICU greater than 24 hours
* Adherence to study

Exclusion Criteria:

* Patients with poor prognosis or palliation;
* Preexisting neuromuscular diseases;
* Immobility or restriction to bed prior to admission;
* Nonunions and amputations;
* Osteomioarticular, cognitive or neurological impairment;
* Non-cooperation;
* Specific contraindications to the application of evaluation methods;
* Hemodynamic or respiratory instability within 48 hours of ICU admission preventing evaluation muscle strength and functional capacity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12; Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Respiratory muscle strength | 48 hours
  Respiratory muscle strength will be assessed through the maximum inspiratory pressure (MIP) and maximal expiratory pressure (MEP).
Peripheral muscle strength | 48 hours
  The peripheral muscle strength will be assessed through the Medical Research Council score (MRC) and hand grip test.
Functional capacity | 48 hours
  The functional capacity will be assessed through the Functional Independence Measure (FIM) and Physical Function ICU Test Score (PFIT-s).

CONTACTS AND LOCATIONS:
Overall Officials: Maria KF Richtrmoc, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Real Hospital Português de Beneficência, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Williams TA, Dobb GJ, Finn JC, Webb SA. Long-term survival from intensive care: a review. Intensive Care Med. 2005 Oct;31(10):1306-15. doi: 10.1007/s00134-005-2744-8. Epub 2005 Aug 24. PMID 16132895
- [Result] Rossi PJ, Edmiston CE Jr. Patient safety in the critical care environment. Surg Clin North Am. 2012 Dec;92(6):1369-86. doi: 10.1016/j.suc.2012.08.007. Epub 2012 Oct 6. PMID 23153874
- [Result] Neideen T. Monitoring devices in the intensive care unit. Surg Clin North Am. 2012 Dec;92(6):1387-402. doi: 10.1016/j.suc.2012.08.010. Epub 2012 Oct 13. PMID 23153875